CLINICAL TRIAL: NCT00683657
Title: A 4-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial To Evaluate The Efficacy And Safety Of Saxagliptin In Comparison To Placebo As Add On Treatment To Metformin XR In Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet And Exercise And A Stable Dose Of Metformin ≥1500 mg/Day
Brief Title: Safety and Efficacy Study of Subjects That Are Taking Saxagliptin Added Onto Metformin XR Compared to Subjects Taking Metformin XR Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-066; Eudract-2008-000976-26
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin 5 mg + Metformin (Experimental)
  Interventions: Drug: Saxagliptin
- Placebo + Metformin (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 5mg, once daily, 4 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin 5 mg + Metformin
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 4 weeks
  Arms: Placebo + Metformin

SUMMARY:
This protocol will compare 24 hour glucose control for subject taking saxagliptin and metformin extended release (XR) versus metformin XR alone

ELIGIBILITY:
Inclusion Criteria:

* ≥18- and ≤77-years-old
* Type 2 diabetes
* Taking metformin immediate release (IR) or XR ≥1500 mg for at least 8 weeks as monotherapy
* Glycosylated hemoglobin (A1C) ≥7% and ≤10%
* Body mass index (BMI) ≤40 kg/m2

Exclusion Criteria:

* Women of childbearing potential unable or unwilling to use acceptable birth control
* Women who are pregnant or breastfeeding
* Significant cardiovascular history
* Active liver disease
* Renal impairment

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (13):
  - Dedicated Phase I, Inc., Phoenix, Arizona
  - Amcr Institute, Inc, Escondido, California
  - Irvine Center For Clinical Research, Inc., Irvine, California
  - Pacific Sleep Medicine Services (Avastra Clinical Trials), Redlands, California
  - Advantage Clinical Research, Santa Ana, California
  - Orange County Research Center, Tustin, California
  - River Birch Research Alliance, Llc, Blue Ridge, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Clinilabs, Inc., New York, New York
  - Covance Cru, Inc., Portland, Oregon
  - Dgd Research, Inc., San Antonio, Texas
  - Avastra Clinical Trials, Midvale, Utah
- Local Institution, Martínez, Buenos Aires, Argentina
- Israel (4):
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Ẕerifin
- Local Institution, Milan, Italy
- Mexico (2):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Monterrey, Nuevo León
- Philippines (2):
  - Local Institution, Cebu City
  - Local Institution, Marikina City
- Local Institution, Ponce, Puerto Rico, Puerto Rico
- Sweden (3):
  - Local Institution, Lund, Sweden
  - Local Institution, Gothenburg
  - Local Institution, Huddinge

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 218 subjects were enrolled and 128 entered the 4-week dietary and exercise, and metformin extended release (XR) lead-in period. Thirty-five subjects did not enter treatment period (21 no longer met study criteria, 7 withdrew consent, 7 for poor protocol compliance).
Groups:
- Saxagliptin 5 mg + Metformin: Saxagliptin tablets, 5 mg, taken orally once daily for 4 weeks, plus metformin XR.
- Placebo + Metformin: Placebo tablets, taken orally once daily for 4 weeks, plus metformin XR.
Period: Overall Study
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Started | 46 | 47
Randomized Subjects Data Set | 46 (Randomized subjects who took at least 1 dose of double-blind study medication.) | 47 (Randomized subjects who took at least 1 dose of double-blind study medication.)
Completed | 45 | 46
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Subject Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.50 (9.20) | 55.77 (9.14) | 55.14 (9.14)
Age, Customized [Number; unit: participants]
  <65 years | 40 | 38 | 78
  >= 65 years to <75 years | 6 | 8 | 14
  >= 75 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 26 | 23 | 49
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 39 | 43 | 82
  Black/African American | 3 | 2 | 5
  Asian | 2 | 1 | 3
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-Hour Mean Weighted Glucose (MWG) at Week 4
Description: Adjusted mean change from baseline in MWG achieved with saxagliptin 5 mg plus metformin XR versus placebo plus metformin XR at Week 24. MWG was calculated as the area under the curve (AUC) for the full 24 hours expressed as average mg/dL. Glucose measurements were collected 30 minutes before and just prior to each meal (0 minutes) and 30, 60, 120, and 180 minutes after each meal (with 1 additional measurement at 240 minutes after the evening meal), midnight, 3 AM, and at end-of-domicile visit 24 hours after the first measurement. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in an analysis of change from baseline to Week 4 the subject must have had a baseline and a Week 4 measurement.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 41 | 44
mg/dL
  Baseline Mean | 177.5 (4.99) | 181.2 (6.30)
  Week 4 Mean | 163.8 (5.09) | 184.2 (7.05)
  Adjusted Mean Change from Baseline | -13.8 (2.99) | 3.0 (2.89)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; With 39 subjects per treatment group, there was a 93% power for the primary endpoint to detect a difference in 24-hour mean weighted glucose of 16 mg/dL between saxagliptin and placebo, assuming a standard deviation of 20 mg/dL. Assuming a dropout rate of 15%, a total of 92 subjects (46 subjects per treatment arm) needed to be randomized; Test type: Superiority or Other; p = 0.0001, ANCOVA — Between-group comparisons significant at alpha = 0.05, significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; ANCOVA Model: post - pre = pre treatment; Mean Difference (Final Values) = -16.8, 95% CI 2-sided [-25.1 to -8.5], Standard Error of Mean 4.16 — Mean difference = adjusted mean change for saxagliptin 5 mg + Metformin - adjusted mean change for Placebo + Metformin

2. Secondary Outcome: Change From Baseline in 4-Hour Mean Weighted Postprandial Plasma Glucose at Week 4
Description: Adjusted mean change from baseline in 4-hour mean weighted postprandial (after mealtime) plasma glucose after the evening meal during 24-hour domicile visits evaluated both at pre-randomization (baseline) and at Week 4. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 40 | 44
mg/dL
  Baseline Mean | 212.1 (6.80) | 211.1 (6.60)
  Week 4 Mean | 181.4 (6.79) | 210.8 (8.02)
  Adjusted Mean Change from Baseline | -30.7 (5.14) | -0.4 (4.90)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model: post - pre = pretreatment; Mean Difference (Final Values) = -30.2, 95% CI 2-sided [-44.4 to -16.1], Standard Error of Mean 7.10 — Mean difference = adjusted mean change for saxagliptin 5 mg + Metformin - adjusted mean change for Placebo + Metformin

3. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose After the Evening Meal at Week 4
Description: Adjusted mean change from baseline in 2-hour postprandial plasma glucose after the evening meal during 24-hour domicile visits, evaluated both at pre-randomization (baseline) and at Week 4. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 41 | 44
mg/dL
  Baseline Mean | 237.6 (8.87) | 233.1 (7.74)
  Week 4 Mean | 198.5 (8.82) | 231.1 (9.22)
  Adjusted Change from Baseline | -38.2 (7.49) | -2.8 (7.23)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model: post - pre = pretreatment; Mean Difference (Final Values) = -35.4, 95% CI 2-sided [-56.2 to -14.7], Standard Error of Mean 10.41 — Mean difference = adjusted mean change for saxagliptin 5 mg + Metformin - adjusted mean change for Placebo + Metformin

4. Secondary Outcome: Change From Baseline in Mean Daily Glucose at Week 4
Description: Adjusted mean change from baseline in daily glucose at Week 4. Mean daily glucose was calculated based on finger stick glucose measurements collected by the subjects at home in a 3-day period, prior to collection of the 24-hour blood samples at baseline and Week 4. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 38 | 44
mg/dL
  Baseline Mean | 179.0 (5.76) | 184.9 (7.14)
  Week 4 Mean | 167.5 (4.87) | 191.8 (8.41)
  Adjusted Change from Baseline | -11.7 (3.02) | 7.0 (2.94)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA Model: post - pre = pretreatment; Mean Difference (Final Values) = -18.7, 95% CI 2-sided [-27.1 to -10.3], Standard Error of Mean 4.22 — Mean difference = adjusted mean change for saxagliptin 5 mg + Metformin - adjusted mean change for Placebo + Metformin

5. Secondary Outcome: Change From Baseline in 2-Day Average Fasting Plasma Glucose (FPG) at Week 4
Description: Adjusted mean change from baseline in 2-day average of FPG at baseline and Week 4. Baseline value=the average of the values at Day -2 and Day 1. Week 4 measurement=average of Day 26 and Day 28 value during the double blind period. At pre-randomization and Day 28 the FPG value was the plasma glucose value collected 30 minutes prior to the morning meal during domicile visits. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 46 | 47
mg/dL
  Baseline Mean | 152.2 (4.14) | 158.9 (5.80)
  Week 4 Last Observation Carried Forward Mean | 141.9 (3.99) | 162.9 (6.00)
  Adjusted Mean Change from Baseline | -10.8 (2.84) | 4.5 (2.81)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA Model: post - pre = pretreatment; Mean Difference (Final Values) = -15.3, 95% CI 2-sided [-23.3 to -7.4], Standard Error of Mean 4.00 — Mean difference = adjusted mean change for saxagliptin 5 mg + Metformin - adjusted mean change for Placebo + Metformin

ADVERSE EVENTS:
Arm/Group | PLACEBO + MET | SAXA 5MG + MET
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 5/47 | 1/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO + MET (N=47) | SAXA 5MG + MET (N=46)
HEADACHE (Nervous system disorders) | 3 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.